CLINICAL TRIAL: NCT07030829
Title: Efficacy and Safety of Laser Versus Electrohydraulic Lithotripsy for Difficult Biliary Stones: A Randomized Controlled Trial
Brief Title: Laser vs Electrohydraulic Lithotripsy for Difficult CBD Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Varayu Prachayakul, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SI 066/2025
Record Dates: First submitted 2025-02-26; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Common Bile Duct Stone
Keywords: Common bile duct stones; CBD stones; Difficult CBD stones; ERCP; Spyglass; Cholangioscopy; Lithrotripsy; Laser lithrotripsy; EHL; Electrohydraulic Lithotripsy
MeSH Terms: conditions — Gallstones | interventions — Lithotripsy, Laser; Lithotripsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser Lithotripsy (Experimental)
  Interventions: Device: Laser Lithotripsy
- Electrohydraulic Lithotripsy (Experimental)
  Interventions: Device: Electrohydraulic Lithotripsy

INTERVENTIONS:
Device: Laser Lithotripsy — Laser Lithotripsy
  Arms: Laser Lithotripsy
Device: Electrohydraulic Lithotripsy — Electrohydraulic Lithotripsy
  Arms: Electrohydraulic Lithotripsy

SUMMARY:
Common bile duct (CBD) stones are a frequent condition that can lead to severe complications if not treated. The standard approach involves endoscopic retrograde cholangiopancreatography (ERCP) with sphincterotomy and stone extraction using balloons or baskets. However, approximately 10-15% of cases involve "difficult CBD stones" that cannot be removed using conventional methods.

According to the European Society of Gastrointestinal Endoscopy (ESGE), difficult CBD stones are characterized by large size (≥15 mm), impaction, multiple stones, difficult locations (e.g., intrahepatic or cystic ducts), or altered anatomy due to previous surgeries. These cases require advanced techniques such as single-operator cholangioscopy (SOC) using the SpyGlass DS system, which allows direct stone visualization and lithotripsy-assisted fragmentation.

Two primary lithotripsy methods are available:

Electrohydraulic Lithotripsy (EHL): Uses shock waves from electrical energy to break stones.

Laser Lithotripsy (LL): Uses laser energy to fragment stones through a water-mediated medium.

While both techniques are effective, studies suggest LL has a higher first-attempt stone clearance rate (82-100%) compared to EHL (70.9-75%). However, EHL is more cost-effective and widely available, whereas LL offers greater precision but at a higher cost. Currently, no randomized controlled trial (RCT) directly compares their efficacy, procedural time, complication rates, or operator satisfaction.

This study aims to fill that gap by conducting a randomized trial comparing EHL and LL in the treatment of difficult CBD stones. The primary outcome is the success rate of complete stone clearance in the first session, while secondary outcomes include procedural duration, post-procedural complications, and operator satisfaction.

The findings will provide critical evidence for optimizing endoscopic stone management, improving patient outcomes, and guiding healthcare resource allocation.

DETAILED DESCRIPTION:
Common bile duct (CBD) stones are a prevalent condition that can lead to severe complications if left untreated. The standard treatment method involves endoscopic retrograde cholangiopancreatography (ERCP) for stone removal. Conventional techniques include sphincterotomy combined with balloon or basket extraction. However, approximately 10-15% of patients present with "difficult CBD stones," which cannot be effectively removed using standard techniques.

The European Society of Gastrointestinal Endoscopy (ESGE) defines difficult CBD stones as those meeting one or more of the following criteria: stone size ≥15 mm, impacted stones, multiple stones, stones in difficult-to-access locations (e.g., intrahepatic or cystic ducts), barrel-shaped stones, or stones in patients with altered anatomy due to prior surgical interventions (e.g., Roux-en-Y reconstruction). These cases often require specialized techniques to achieve successful stone clearance while minimizing complications.

Intervention and Rationale:

Single-operator cholangioscopy using the SpyGlass system has become a widely adopted approach for managing difficult CBD stones. This technique enables direct visualization of the stone and facilitates lithotripsy, which fragments stones into smaller pieces for easier removal. The two primary lithotripsy techniques available are:

Electrohydraulic Lithotripsy (EHL): Uses shock waves generated by electrical energy transmitted through a probe to fragment stones.

Laser Lithotripsy (LL): Uses laser energy delivered through a water-mediated medium to break stones into smaller pieces.

Both techniques have demonstrated high success rates in stone fragmentation and removal, but debate persists regarding their relative efficacy. Some studies suggest that LL achieves higher first-attempt stone clearance rates (82-100%) compared to EHL (70.9-75%). However, EHL is generally more cost-effective and widely available, whereas LL offers greater precision at a higher procedural cost.

Objective:

This study aims to compare the effectiveness of EHL and LL in the management of difficult CBD stones through a randomized controlled trial (RCT). The primary outcome is the success rate of complete stone clearance in the first session. Secondary outcomes include procedural time, complication rates, and operator satisfaction.

Study Design:

Study Type: Randomized Controlled Trial

Study Population: Patients diagnosed with difficult CBD stones requiring lithotripsy

Intervention Groups:

Group 1: EHL via SpyGlass DS

Group 2: LL via SpyGlass DS

Primary Endpoint: First-session complete stone clearance rate

Secondary Endpoints:

Procedural duration

Post-procedural complications

Operator satisfaction

Significance:

The findings from this study will provide valuable evidence for endoscopists regarding the optimal lithotripsy method for difficult CBD stones, ultimately improving patient outcomes and healthcare resource utilization. By identifying the most effective and efficient technique, this study aims to optimize treatment strategies and enhance clinical decision-making in endoscopic stone management.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Difficult CBD stone
* Large CBD stone (stone > 1.5 cm) or Stone impaction or CBD stones that were not completely removed using conventional techniques.

Exclusion Criteria:

* Pregnancy
* Unstable vital signs
* Severe comorbidities
* Uncorrected coagulopathy
* Surgically altered anatomy
* Unable to complete informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Electrohydraulic Lithotripsy (EHL) and Laser Lithotripsy (LL) | During the procedure
  Comparison of the effectiveness of Electrohydraulic Lithotripsy (EHL) and Laser Lithotripsy (LL) by examining the success rate of complete stone removal on the first procedure.

SECONDARY OUTCOMES:
Procedure time | Periprocedural (Total procedure time usually 1-2 hours)
  Procedure time of ERCP with spyglass
Number of catheters used | Periprocedural
  Number of catheters used
Physician satisfaction | Periprocedural
  Physician satisfaction of EHL vs LL based on questionaire on a scale of 0-5 for ease of use and lithotripsy effect
Procedure-related adverse events | up to 2 weeks after the procedure
  Procedure-related adverse events
Length of hospital stay | through after procedure average 1-2 weeks
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Varayu Prachayakul, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
We are willing to provide our data to researchers who require it. For example, those who want to do systematic review and meta-analysis.
Supporting Information: Study Protocol
Time Frame: Other researchers can contact us anytime.
Access Criteria: We will provide our protocol and/or data upon request.